CLINICAL TRIAL: NCT02559375
Title: PAIN-LESS: Understanding and Alleviating Pain for Cancer Patients in Academic and Community Hospitals
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 26914
Record Dates: First submitted 2015-06-23; First posted 2015-09-24 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Survey

SUMMARY:
This study will increase knowledge of patient preferences for pain treatments, and improve the ability to meet patients pain management needs. This study will assess patient attitudes towards underutilized treatments and identify technologies to increase awareness of such treatments. This study also demonstrate the feasibility of using the Penn Cancer Network in future clinical and cancer control research and better understand how to effectively raise patients awareness of supportive cancer services.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older; Have a primary diagnosis of cancer;
* Have a Karnofsky functional score of 60 or greater (i.e. ambulatory);
* Understand written English;
* Verbally indicate to the RA/RN that they feel physically well enough to complete a survey at the time of approach;
* Report experiencing nonzero pain (on a scale of 0-10) in the last seven days

Exclusion Criteria:

* An inability to understand the requirements of the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Patients
Sampling Method: Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects providing completed surveys | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States